CLINICAL TRIAL: NCT05423860
Title: This is a Human Analytics Longitudinal Observational (HALO) Study. A Phase I Study to Analyze All Available Biomarkers and Determinants of Health to Increase Diagnostic Accuracy While Reducing the Time to Diagnosis of Disease.
Brief Title: Phase I Human Analytics (HALO) Study
Acronym: HALO
Status: Recruiting | Type: Observational
Sponsor: HALO Diagnostics (Industry)
Collaborators: HALO Affiliate Sites (Unknown)
Responsible Party: Sponsor
Other Study IDs: HALO Dx 001; WIRB Pr. No.: 20213955 (Other: WIRB Copernicus Group (WCG))
Record Dates: First submitted 2022-04-29; First posted 2022-06-21 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Cardiovascular Diseases; Cancer; Dementia; Traumatic Brain Injury
Keywords: brain; breast; prostate; cardiac; cancer
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Dementia; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- dementia: Patients with a diagnosis of dementia
  Interventions: Other: no interventions will be performed (observational)
- Prostate cancer: patients with a diagnosis of prostate cancer
  Interventions: Other: no interventions will be performed (observational)
- breast cancer: Patients with a diagnosis of breast cancer
  Interventions: Other: no interventions will be performed (observational)
- Normal: Patients without a diagnosis
  Interventions: Other: no interventions will be performed (observational)
- tramatic brain injury: patients with a diagnosis of traumatic brain injury
  Interventions: Other: no interventions will be performed (observational)

INTERVENTIONS:
Other: no interventions will be performed (observational) — Not applicable. (no interventions will be performed with this observational study

SUMMARY:
Discover, optimize, standardize, and validate clinical-trial measures and biomarkers used to diagnose and differentiate cardiovascular, oncologic, neurologic, and other diseases and disorders. Specifically, our research study endeavors to improve disease and disorder diagnosis to the earliest clinical states, in preclinical states, and to develop ensemble multivariate biomarker risk scores leading to cardiovascular, oncologic, neurologic, and other diseases and disorders.

Additionally, the study aims to:

* Evaluate data analysis techniques to improve diagnostic accuracy and reduce time to diagnosis.
* Evaluate data analysis techniques to improve risk stratification for participants through machine learning algorithms.
* Direct participants to relevant and applicable clinical trials.

DETAILED DESCRIPTION:
Electronic medical records contain data that may indicate increased risk for certain diseases and disorders, but clinicians cannot easily discern the subtle patterns required to change their diagnostic and treatment patterns. This study seeks to use machine learning and data analysis techniques to increase diagnostic confidence and reduce time-to-diagnosis related to cardiovascular, oncologic, neurologic, and other diseases and disorders.

The study endeavors to develop ensemble multivariate biomarker risk scores to predict future development of diseases and disorders, improve diagnosis in preclinical states and increase diagnostic accuracy in the earliest clinical states. We also aim to evaluate data analysis techniques to improve diagnostic accuracy and reduce time to diagnosis, improve risk stratification for participants through machine learning algorithms and direct participants to relevant and applicable clinical trials upon physician review, approval and recommendation.

ELIGIBILITY:
Inclusion Criteria:

Treatment Naïve patients:

* Male, 45 years of age or older.
* Diagnosis of prostate adenocarcinoma.
* Clinical stage T1c or T2a.
* Gleason score of 7 (3+4 or 4+3) or less.
* Three or fewer biopsy cores with prostate cancer.
* PSA density not exceeding 0.375.
* One, two, or three tumor suspicious regions identified on multiparametric MRI.
* Negative radiographic indication of extra-capsular extent.
* Karnofsky performance status of at least 70.
* Estimated survival of 5 years or greater, as determined by treating physician.
* Tolerance for anesthesia/sedation.
* Ability to give informed consent.
* At least 6 weeks since any previous prostate biopsy.
* MR-guided biopsy confirmation of one or more MRI-visible prostate lesion(s) with Gleason score of 7 (3+4 or 4+3) or less.

Salvage candidates will be accepted upon physician referral.

Exclusion Criteria:

* Presence of any condition (e.g., metal implant, shrapnel) not compatible with MRI.
* Severe lower urinary tract symptoms as measured by an International Prostate Symptom Score (IPSS) of 20 or greater
* History of other primary non-skin malignancy within previous three years.
* Diabetes
* Smoker

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2037-03 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer Gleason score | Up to 5 years after treatment
  Measure a patient's prostate cancer Gleason score for patients with a prostate cancer diagnosis and record the measurement again at 3, 6, 9 months and annually for 5 years after treatment. We will use the pathology report submitted by the pathologist. The Gleason Score ranges from 1-5 and describes how much the cancer from a biopsy looks like healthy tissue (lower score) or abnormal tissue (higher score).
Prostate cancer ISUP grade group | Up to 5 years after treatment
  Measure a patient's prostate cancer ISUP grade group for patients with a prostate cancer diagnosis and record the measurement again at 3, 6, 9 months and annually for 5 years after treatment. We will use the pathology report submitted by the pathologist. The International Society of Urological Pathology (ISUP) guidelines grades the cancer between 1 and 5 depending on the Gleason score. The lower the grade the less likely the cancer is to spread.
Prostate cancer staging parameters | Up to 5 years after treatment
  TNM stage and metastasis-free survival, documentation of tumor, lymph node and osseous involvement
Prostate cancer specific mortality | Up to 5 years
  Proportion of men who expire directly due to prostate cancer

SECONDARY OUTCOMES:
Lower urinary tract symptoms (LUTS) | Up to 5 years after treatment
  Measure patient's prostate symptom score for patients with a prostate cancer diagnosis and repeat the survey at 3, 6, 9 months and annually for 5 years after treatment. We will use the International Prostate Symptom Score (I-PSS) survey. The International Prostate Symptom Score (IPSS) is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia (BPH).
Erectile function | Up to 5 years after treatment
  Measure a patient's sexual health score for patients with a prostate cancer diagnosis and repeat the survey at 3, 6, 9 months and annually for 5 years after treatment. We will use the Sexual Health Inventory for Men survey. The Sexual Health Inventory for Men (SHIM) is a widely used scale for screening and diagnosis of erectile dysfunction (ED) and severity of ED in clinical practice and research.
Emotional well-being | Up to 5 years after treatment
  Measure a patient's level of distress for patients with a prostate cancer diagnosis and repeat the survey at 3, 6, 9 months and annually for 5 years after treatment. We will use the NCCN-DT survey. The NCCN Distress Thermometer and Problem List is a well-known screening tool among cancer care providers. The survey is a one-item, 11-point Likert scale represented on a visual graphic of a thermometer that ranges from 0 (no distress) to 10 (extreme distress), with which patients indicate their level of distress over the course of the week prior to assessment.
Incontinence level | Up to 5 years after treatment
  Measure a patient's incontinence for patients with a prostate cancer diagnosis and repeat the survey at 3, 6, 9 months and annually for 5 years after treatment. We will use the ICIQ-UI Short Form survey. The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world.
PI-RADS category | Up to 5 years after treatment
  Measure a patient's PI-RADS category for patients with a prostate cancer diagnosis and record measurement again at 3, 6, 9 months and annually for 5 years after treatment. We will use the radiology report submitted by the radiologist. Radiologists use the Prostate Imaging Reporting and Data System (PI-RADS) to report how likely it is that a suspicious area is a clinically significant cancer. In the PI-RADS scale, each lesion is assigned a score from 1 to 5 indicating the likelihood of clinically significant cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Hancock, MD, Principal Investigator — HALO Diagnostics; Erik W. Peterson, BS, Study Director — HALO Diagnostics
Locations (1):
- Desert Medical Imaging, Indian Wells, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication
Time Frame: Interval updates may be presented at scientific meetings as available. Interim results may also be published.
Access Criteria: Scientists and physicians

REFERENCES:
- [Background] Weng SF, Reps J, Kai J, Garibaldi JM, Qureshi N. Can machine-learning improve cardiovascular risk prediction using routine clinical data? PLoS One. 2017 Apr 4;12(4):e0174944. doi: 10.1371/journal.pone.0174944. eCollection 2017. PMID 28376093
- [Background] Wang X, Oldani MJ, Zhao X, Huang X, Qian D. A review of cancer risk prediction models with genetic variants. Cancer Inform. 2014 Sep 21;13(Suppl 2):19-28. doi: 10.4137/CIN.S13788. eCollection 2014. PMID 25288876
- See also: HALO Diagnostics — http://www.halodx.com